CLINICAL TRIAL: NCT01672203
Title: Incidence of CTEPH in Dependence of Thrombus Location in Patients With Acute Pulmonary Embolism and Index Fibrinolysis
Brief Title: Chronic Thromboembolic Pulmonary Hypertension (CTEPH) Incidence in Patients With Central Versus Peripheral Embolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Fikret Er, MD, University of Cologne
Other Study IDs: UKK-PostLE
Record Dates: First submitted 2012-08-15; First posted 2012-08-24 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: CTEPH

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- PE peripheral with fibrinolysis: Patients with peripheral PE who received fibrinolysis therapy
- PE peripheral, no fibrinolysis: Patients with peripheral PE who did not receive fibrinolysis
- PE central with fibrinolysis: Patients with central PE who received fibrinolysis therapy
- PE central, no fibrinolysis: Patients with central PE who did not receive fibrinolysis

SUMMARY:
Chronic thromboembolic pulmonary hypertension (CTEPH) has been associated with increased morbidity and mortality. Patients with pulmonary embolism (PE) have elevated risk for development of CTEPH. It is not known, whether the location of pulmonary embolism (central vs. peripheral) nor fibrinolysis have an impact of CTEPH incidence. This study has been performed to assess the CTEPH incidence in different populations: in patients with central vs. peripheral PE and in patients with or without fibrinolysis therapy for PE.

DETAILED DESCRIPTION:
The embolus localization during index pulmonary embolism might be of potential relevance for CTEPH development.

In the present study patients with confirmed pulmonary embolism for at least 12 months will be screened for CTEPH. The incidence of CTEPH will be correlated to thrombus location (central vs. peripheral) and the index use of fibrinolysis.

ELIGIBILITY:
Inclusion Criteria:

* acute pulmonary embolism for at least 12 months

Exclusion Criteria:

* known pulmonary hypertension other than CTEPH

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalized for acute pulmonary embolism at the University Hospital of Cologne.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
CTEPH | participants will be followed at least one year after acute pulmonary embolism, an expected average of 5 years follow-up is estimated
  Incidence of CTEPH

CONTACTS AND LOCATIONS:
Overall Officials: Fikret Er, MD, Principal Investigator — University of Cologne
Locations (1):
- Heart Center of the University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany